CLINICAL TRIAL: NCT03209674
Title: Registry for the Improvement of Postoperative OutcomeS in Cardiac and Thoracic surgEry
Acronym: RIPOSTE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Other Study IDs: RIPOSTE
Record Dates: First submitted 2017-07-03; First posted 2017-07-06 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-01

CONDITIONS: Heart Diseases; Death; Postoperative Complications; Cardiac Complication
Keywords: Cardiac surgery; Thoracic surgery
MeSH Terms: conditions — Heart Diseases; Death; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cardiothoracic surgery — Cardiac or thoracic procedure

SUMMARY:
The registry for the improvement of postoperative outcomes in cardiac and thoracic surgery aims to prospectively collect data in order to test the association between various preoperative and per-operative variables ; and several postoperative outcomes such as mortality, shock, redo surgery, sepsis and extracorporeal life-support.

DETAILED DESCRIPTION:
Cardiac and thoracic surgery is plagued by severe morbidity and mortality. Understanding and being able to predict postoperative outcomes may allow to better fit peri-operative care of cardio-thoracic patients.

RIPOSTE database aims to prospectively collect baseline characteristics and per-operative information in order to test associations with the incidence of postoperative outcomes.

Baseline characteristics include: age, EuroSCORE 2 and its components (age, gender, New York Heart Association (NYHA) functional class, angina symptoms, insulin-dependent diabetes mellitus, extracardiac arteriopathy, chronic pulmonary dysfunction, neurological or musculoskeletal dysfunction severely affecting mobility, previous cardiac surgery, renal function with creatinin clearance, active endocarditis, critical preoperative state, left ventricle ejection fraction, recent myocardial infarction, pulmonary artery systolic pressure, procedure urgency and weight of the procedure (coronary artery bypass graft, valve surgery and/or thoracic aorta)) weight, height, preoperative biology and preoperative echocardiography parameters when measured.

Peroperative information include: cardiac bypass duration, type of procedure, implanted device, valve size.

Postoperative outcomes include: death, postoperative shock, mediastinitis, length of stay in intensive care unit, overall length of stay, blood transfusion.

ELIGIBILITY:
Inclusion Criteria:

* all patients eligible for cardiac or thoracic surgery

Exclusion Criteria:

* non applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing cardiac or thoracic surgery in CMC Ambroise Paré
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | During follow-up, until discharge from hospital, up to 1 year.
  death occurring in the same hospital where the operation took place before discharge from the hospital

SECONDARY OUTCOMES:
Postoperative shock | In the first 24 hours after surgery
  Use of catecholamines (dobutamine, norepinephrine and/or epinephrine) in order to achieve adequate cardiac output (cardiac index > 2.2 l/min/m2), in the first 24 hours after surgery
Length of stay in the ICU (days) | During follow-up, until discharge from the ICU, up to 1 year.
  length of stay in the intensive care unit after cardiac or thoracic surgery
Total length of stay (days) | During follow-up, until discharge from the hospital, up to 1 year.
  length of stay in the hospital, including preoperative period
Mediastinitis | During follow-up, until discharge from the hospital, up to 1 year.
  Incidence of mediastinitis in the postoperative period
Redo surgery | During follow-up, until discharge from the hospital, up to 1 year.
  Redo surgery after primary surgery
Pneumoniae | During follow-up, until discharge from the hospital, up to 1 year.
  Hospital-acquired or Ventilator-acquired pneumonia as defined by Center for Disease Control guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Caroline Merand, Study Chair — CMC Ambroise Paré
Locations (1):
- CMC Ambroise Paré, Neuilly-sur-Seine, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No
non-applicable.

REFERENCES:
- [Derived] Suc G, Estagnasie P, Brusset A, Procopi N, Squara P, Nguyen LS. Effect of BNP on risk assessment in cardiac surgery patients, in addition to EuroScore II. Sci Rep. 2020 Jul 2;10(1):10865. doi: 10.1038/s41598-020-67607-0. PMID 32616802